CLINICAL TRIAL: NCT00947596
Title: Development of an Inhaled, Dry Powder Delivery System for the Administration of Atropine Sulfate
Brief Title: A Study of Inhaled Atropine Sulfate in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicroDose Defense Products L.L.C. (Industry)
Collaborators: University of Pittsburgh (Other); U.S. Army Space and Missile Defense Command (U.S. Federal Agency)
Responsible Party: Michael Donahoe, MD, University of Pittsburgh Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PRO07030057
Record Dates: First submitted 2009-07-22; First posted 2009-07-28 (Estimated); Last update posted 2010-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Organophosphorus Poisoning
Keywords: Atropine; Aerosol; Inhaler; Dry Powder
MeSH Terms: conditions — Organophosphate Poisoning | interventions — Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atropine Dry Powder Inhaler (Experimental)
  Interventions: Drug: atropine sulfate
- Atropen Autoinjector (Active Comparator)
  Interventions: Drug: atropine sulfate

INTERVENTIONS:
Drug: atropine sulfate — dry powder for inhalation
  Other Names: MicroDose inhaler
  Arms: Atropine Dry Powder Inhaler
Drug: atropine sulfate — intramuscular injection
  Arms: Atropen Autoinjector

SUMMARY:
MicroDose Defense Products, LLC is developing an atropine dry powder inhaler (ADPI). This pilot study compares the pharmacokinetics (PK) of inhaled dry powder atropine as delivered by the ADPI to atropine delivery from the AtroPen autoinjector.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 18-55 years of age.
* Subjects will be able to read and comprehend the English language.

Exclusion Criteria:

* Subjects weighing less than 100 lbs.
* Women of childbearing potential who are pregnant or unwilling to undergo pregnancy testing; females with positive pregnancy testing on either screening day or any test day will be excluded. Nursing mothers will be excluded
* Persons unable or unwilling to complete written informed consent (No proxy consent will be obtained).
* Persons with a past medical history or symptoms of pulmonary disease (including but not limited to: asthma, COPD, Emphysema, Sarcoidosis, Lung Cancer, Pulmonary Embolism, Pulmonary Hypertension))or cardiac disease (coronary artery disease, hypertension, angina, arrhythmias, palpitations, past myocardial infarction history).
* Persons with a previous history or symptoms of adverse reaction to atropine.
* Persons with history or symptoms of prostate hypertrophy or prostate cancer.
* Persons with a history or symptoms of pyloric stenosis.
* Persons with a history or symptoms of high blood pressure or a diagnosis of cerebral vascular accident (CVA) or transient ischemic attack (TIA).
* Subjects with a history or symptoms of urological disorders or renal insufficiency.
* Subjects with a history or symptoms of diabetes.
* Persons demonstrating increased intraocular pressure, an abnormal optical exam, or history of glaucoma.
* Persons demonstrating a one second forced expiratory volume (FEV1) or a forced vital capacity (FVC) of less than 70% of predicted either at screening or during pre test exam will be excluded
* Persons demonstrating any kind of irregular heart rhythm during pre test screening will be excluded. Persons demonstrating any irregular rhythms during testing will be immediately removed.

from testing and receive appropriate care and referral from the study physician

* Persons will be excluded if any two laboratory tests characterizing a specific organ system are more than 10% outside of normal range
* Subjects with screening day vital signs considered to be beyond normal range will be excluded. This will include BP systolic > 140, Diastolic > 90, HR > 100, RR > 20, temp > 38.
* The study physician will have the discretion to exclude subjects that he/she feels will not be able to safely able to participate in these studies based on review of all screening materials.
* Self reported tobacco use or positive cotinine testing.
* Any individuals with positive results on a urine drug screening will be excluded.
* Persons with an O2 saturation value < 92%.
* Persons who have performed other medical studies involving drug delivery in the last 30 days.
* Blood donation in the last 30 days.
* Subjects regularly utilizing any of the following medications will be excluded: amantadine, quinidine, phenothiazines, tricyclic antidepressants, digoxin, potassium chloride and potassium citrate formulations, topiramate, zonisamide.
* Subjects under 18 years of age.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To characterize pharmacokinetic endpoints for atropine dry powder inhalation (Cmax, Tmax, AUC) and compare these to intramuscular pharmacokinetics (Atropen autoinjector) | Multiple plasma samples collected up to 12 hours post dose

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of atropine dry powder inhalation (Clinical Labs testing, Pulse, Pulse Oximetry, Temperature, Heart Rate, Pulmonary Function Tests, Respiratory Rate, Near Point of Accommodation, Pupil Size). | up to 36 days (including 14 day screening period)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donahoe, M.D., Principal Investigator — Division of Pulmonary, Allergy and Critical Care Medicine, University of Pittsburgh; Timothy Corcoran, Ph.D., Study Director — Division of Pulmonary, Allergy and Critical Care Medicine, University of Pittsburgh
Locations (1):
- Montefiore Hospital Clinical and Translational Research Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- See also: Product Description — http://mdtx.com/pipeline/proprietary-products/atropine/